CLINICAL TRIAL: NCT01105091
Title: A Phase IV, Open-label, Randomized, Multicenter Study of the Safety, Tolerability,and Pharmacokinetics of ACT- 385781A Compared to Flolan® in Injectable Prostanoid Treatment-naïve Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Epoprostenol for Injection in Pulmonary Arterial Hypertension
Acronym: EPITOME-1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AC-066A401
Record Dates: First submitted 2010-04-15; First posted 2010-04-16 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; PAH; EPITOME-1
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ACT-385781A (Actelion Epoprostenol)
  Interventions: Drug: ACT-385781A (Actelion Epoprostenol)
- 2 (Active Comparator): Flolan®
  Interventions: Drug: Flolan®

INTERVENTIONS:
Drug: ACT-385781A (Actelion Epoprostenol) — per Prescribing Information
  Arms: 1
Drug: Flolan® — Per Prescribing Information
  Arms: 2

SUMMARY:
This is a prospective, multi-center, open-label, randomized, Phase IV exploratory study comparing safety, tolerability, pharmacokinetics, and effectiveness of ACT-385781A and Flolan (epoprostenol sodium) in patients with pulmonary arterial hypertension who are naïve to injectable prostanoid treatment and in need of such treatment. Approximately 30 patients from 8 U.S. clinical sites will be randomized to receive either ACT-385781A or Flolan (2:1 respectively) for 28 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-65 years
2. Patients with the following types of pulmonary arterial hypertension (PAH) belonging to WHO Group I:

   * Idiopathic (IPAH)
   * Heritable (HPAH)
   * Associated (APAH) with

     * Connective tissue diseases
     * Drugs and toxins
3. Patients with PAH in modified NYHA functional class III or IV at the time of enrollment in need of injectable epoprostenol.
4. Patients must be injectable prostanoid treatment-naïve and either

   * newly diagnosed and not yet treated with specific PAH therapies or
   * currently treated with existing background PAH therapy with one or more of the following medications for 90 days prior to enrollment and on a stable dose for 30 days prior to enrollment:

     * Bosentan
     * Ambrisentan
     * Sildenafil
     * Tadalafil
5. Women of childbearing potential must use a reliable method of contraception.

Exclusion Criteria:

1. Patients with respiratory and/or cardiovascular distress in need of emergency care including i.v. epoprostenol administration or any vasopressive i.v. drugs
2. Known pulmonary veno-occlusive disease (PVOD)
3. Current use of i.v. inotropic agents
4. Tachycardia with heart rate > 120 beats/min
5. Pulmonary arterial hypertension related to any condition other than those specified in the inclusion criteria
6. Known hypersensitivity to the formulations of ACT-385781A or any of its excipients, and Flolan or any of its excipients
7. Use of inhaled iloprost or treprostinil during the week prior to screening
8. Cerebrovascular events (e.g., transient ischemic attack or stroke) within 6 months of screening
9. History of myocardial infarction
10. History of left-sided heart disease, including any of the following:

    * hemodynamically significant aortic or mitral valve disease
    * restrictive or congestive cardiomyopathy
    * left ventricular ejection fraction < 40% by multigated radionucleotide angiogram(MUGA),angiography, or echocardiography
    * unstable angina pectoris
    * life-threatening cardiac arrhythmias
11. Chronic bleeding disorder
12. Infection(s) within the past month that in the mind of the investigator would contraindicate the use of epoprostenol
13. Pregnancy or breast-feeding
14. Participation in another clinical trial, except observational (noninterventional), or receipt of an investigational product within 30 days prior to randomization
15. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease
16. Known concomitant life-threatening disease other than PAH with a life expectancy < 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Benton, PharmD, Study Director — Actelion

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at seven Pulmonary Hypertension centers in the U.S. Patients were recruited from these Pulmonary Hypertension medical clinics. Recruitment period was March 2010 through March 2011.
Pre-assignment Details: Up to 14 days screening period.
Groups:
- ACT-385781A (Epoprostenol for Injection): The prepared solution was administered by continuous intravenous (i.v.) infusion via a central venous catheter using an ambulatory infusion pump. Administration was to be initiated at an infusion rate of 2 ng/kg/min, with up titration according to therapeutic need and tolerability.
- Flolan® (Epoprostenol Sodium) for Injection: The prepared solution was administered by continuous i.v. infusion via a central venous catheter using an ambulatory infusion pump. Administration was to be initiated at an infusion rate of 2 ng/kg/min, with up titration according to therapeutic need and tolerability
Period: Overall Study
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Started | 20 | 10
Completed | 18 | 10
Not Completed | 2 | 0
Not completed — Death | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 10 | 28
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.0 (17.0) | 44.1 (12.6) | 44.7 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 6 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 20 | 10 | 30
New York Heart Association (NYHA) Functional Class [Number; unit: participants] — Disease severity was assessed by NYHA classification of PH criteria: Class I: no limitation of physical activity (PA). Ordinary PA: no undue dyspnea/fatigue, chest pain, near syncope. Class II: slight limitation of PA. Comfortable at rest. Ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class III: marked limitation of PA. Comfortable at rest. Less than ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class IV: inability to carry out PA without symptoms. Right heart failure. Dyspnea/fatigue may even have been present at rest. Discomfort increased by any PA.
  participants
    Class I | 0 | 0 | 0
    Class II | 0 | 0 | 0
    Class III | 17 | 8 | 25
    Class IV | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Dose Normalized Pharmacokinetics of 6,15-diketo-13,14-dihydro-Prostacyclin F1alpha at 2 ng/kg/Min
Description: The plasma concentration for the epoprostenol metabolite 6,15-diketo-13,14-dihydro-Prostacyclin F1alpha was measured at 2 ng/kg/min just prior to the next up-titration. Dose-normalized concentrations are used to summarize the results.
Time Frame: Day 1
Population: A per-protocol analysis set that included all patients in the treated set who did not violate the protocol in a way that might affect the evaluation of the effect of the study drug(s) on the pharmacokinetic endpoints.
Measure: Median (Full Range); unit: (pg/ml)/(ng/kg/min)
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 15 | 6
(pg/ml)/(ng/kg/min) | 98.0 [12.5 to 416.5] | 83.1 [36.0 to 158.5]

2. Primary Outcome: Dose Normalized Pharmacokinetics of 6,15-diketo-13,14-dihydro-Prostacyclin F1alpha at 4 ng/kg/Min
Description: The plasma concentration for the epoprostenol metabolite 6,15-diketo-13,14-dihydro-Prostacyclin F1alpha was measured at 4 ng/kg/min just prior to the next up-titration. Dose-normalized concentrations are used to summarize the results.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: (pg/ml)/(ng/kg/min)
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 10 | 6
(pg/ml)/(ng/kg/min) | 90.9 [29.3 to 195.0] | 59.6 [24.9 to 170.5]

3. Primary Outcome: Dose Normalized Pharmacokinetics of 6-keto-Prostacyclin F1alpha at 2 ng/kg/Min
Description: The plasma concentration for the epoprostenol metabolite 6-keto-Prostacyclin F1alpha was measured at 2 ng/kg/min just prior to the next up-titration. Dose-normalized concentrations are used to summarize the results.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: (pg/ml)/(ng/kg/min)
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 15 | 6
(pg/ml)/(ng/kg/min) | 85.5 [12.5 to 374.5] | 109.2 [38.4 to 152.0]

4. Primary Outcome: Dose Normalized Pharmacokinetics of 6-keto-Prostacyclin F1alpha at 4 ng/kg/Min
Description: The plasma concentration for the epoprostenol metabolite 6-keto-Prostacyclin F1alpha was measured at 4 ng/kg/min just prior to the next up-titration. Dose-normalized concentrations are used to summarize the results.
Time Frame: Day 1
Population: as for outcome 1
Measure: Median (Full Range); unit: (pg/ml)/(ng/kg/min)
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 10 | 6
(pg/ml)/(ng/kg/min) | 93.1 [29.8 to 457.5] | 95.0 [33.3 to 201.0]

5. Primary Outcome: Six-minute Walk Distance (6MWD) - Baseline and Day 28
Description: The 6-minute walk test (6MWT) was to be performed prior to initiating study treatment either during the screening visit or on Day 1 prior to drug initiation, and Day 28 (End of treatment (EOT)). This assessment is a non-encouraged test that measures the distance walked for a duration of 6 minutes. The 6MWD was recorded in the Case Report Form (CRF).
Time Frame: Baseline and 28 days (+3 days)
Population: Patients who had both baseline and Day 28 assessments were included in the analysis. The analysis was conducted without replacement of missing values.
Measure: Median (Full Range); unit: meters
Groups:
- ACT-385781A (Epoprostenol for Injection); Flolan (Epoprostenol Sodium) for Injection: The prepared solution was administered by continuous i.v. infusion via a central venous catheter using an ambulatory infusion pump. Administration was to be initiated at an infusion rate of 2 ng/kg/min, with up titration according to therapeutic need and tolerability.
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 17 | 10
meters
  Baseline | 339.0 (84) [45 to 465] | 302.5 (58.8) [25 to 413]
  Day 28 | 288.0 [114 to 506] | 323.5 [90 to 429]

6. Primary Outcome: Patients With New York Heart Association (NYHA) Functional Class Change (Improved or Worsened) From Baseline to Day 28
Description: Disease severity was assessed by NYHA classification of PAH criteria: Class I: no limitation of physical activity (PA). Ordinary PA: no undue dyspnea/fatigue, chest pain, near syncope. Class II: slight limitation of PA. Comfortable at rest. Ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class III: marked limitation of PA. Comfortable at rest. Less than ordinary PA: undue dyspnea/fatigue, chest pain, near syncope. Class IV: inability to carry out PA without symptoms. Right heart failure. Dyspnea/fatigue may even have been present at rest. Discomfort increased by any PA.
Time Frame: From baseline to 28 days (+3 days)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 18 | 10
participants
  Improved Patients | 6 | 3
  Worsened Patients | 0 | 0

7. Primary Outcome: Percentage Central Venous Blood Oxygen Saturation (ScVO2) - Baseline and Day 28
Description: Central venous blood oxygen saturation assessment was performed only in specific centers. Measurements for ScVO2 were performed during the inpatient hospitalization period on Day 1 (prior to drug initiation) and on Day 28 (EOT). Samples for ScVO2 were obtained by aspirating blood from the indwelling central venous catheter. After the sample had been drawn, the catheter was primed with study drug in order to refill the lumen to avoid interruption in treatment and sudden decompensation.
Time Frame: Baseline and 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: percentage oxygen saturation
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 11 | 6
percentage oxygen saturation
  Baseline | 63.0 [55 to 78] | 61.5 [41 to 65]
  Day 28 | 58.0 [36 to 73] | 56.0 [50 to 64]

8. Primary Outcome: Blood Pressure - Baseline and Day 28
Description: Blood pressure (systolic and diastolic) were measured indirectly using an automatic oscillometric device, on the same arm for each measurement. The Blood Pressure was assessed at baseline and at Day 28 (End of Study Treatment visit).
Time Frame: Baseline and 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: mm Hg
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 18 | 10
mm Hg
  Systolic Blood Pressure (Baseline) | 106.5 [81 to 138] | 106.5 [79 to 142]
  Systolic Blood Pressure (Day 28) | 117.5 [98 to 140] | 116.0 [80 to 136]
  Diastolic Blood Pressure (Baseline) | 62.0 [44 to 98] | 68.0 [58 to 99]
  Diastolic Blood Pressure (Day 28)) | 71.0 [62 to 84] | 73.0 [60 to 107]

9. Primary Outcome: Heart Rate - Baseline and Day 28
Description: Heart rate was measured indirectly using an automatic oscillometric device, on the same arm for each measurement. The Heart Rate was assessed at Baseline and at Day 28 (End of Study Treatment visit).
Time Frame: Baseline and 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: Beats per minute
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 18 | 10
Beats per minute
  Baseline | 83.0 [61 to 104] | 77.5 [60 to 105]
  Day 28 | 85.0 [62 to 150] | 88.0 [76 to 112]

10. Primary Outcome: Body Weight - Baseline and Day 28
Description: Body weight was measured both at baseline and day 28.
Time Frame: Baseline and 28 days
Population: as for outcome 5
Measure: Median (Full Range); unit: kg
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Number analyzed (Participants) | 18 | 10
kg
  Baseline | 74.1 [54 to 111] | 74.2 [58 to 103]
  Day 28 | 73.6 [54 to 102] | 73.3 [56 to 99]

ADVERSE EVENTS:
Time Frame: Screening to day 28 for treatment-emergent (TE) adverse events (AEs) during dosing inpatient hospitalization and during outpatient period up to day 28 (EOT). TE serious AEs (SAEs) up to 30 days post study drug.
Description: The assessment of safety was based on the collection of AEs, including SAEs and AEs that resulted in discontinuation of study treatment. All AEs that occurred up to the end of the last day of study treatment were recorded in the CRF and included in the clinical database. SAEs and deaths that occurred up to 30 days after the end of study treatment.
Arm/Group | ACT-385781A (Epoprostenol for Injection) | Flolan® (Epoprostenol Sodium) for Injection
Serious Adverse Events (participants affected / at risk) | 6/20 | 2/10
Other Adverse Events (participants affected / at risk) | 20/20 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | ACT-385781A (Epoprostenol for Injection) (N=20) | Flolan® (Epoprostenol Sodium) for Injection (N=10)
Ascites (Hepatobiliary disorders) | 0/0 (0) | 1 (1) — 34 year female, Flolan, resolved without sequelae / unrelated to Flolan
Cardiac arrest (Cardiac disorders) | 1 (1) | 0/0 (0) — 64 year male, Death (outcome), unrelated to ACT-385781
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Device Related Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Fluid Overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Right Ventricular Failure (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACT-385781A (Epoprostenol for Injection) (N=20) | Flolan® (Epoprostenol Sodium) for Injection (N=10)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse Drug Reaction (General disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Application Site Pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site Hypersensitivity (General disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Catheter Site Discharge (General disorders) | 1 (1) | 0 (0)
Catheter Site Pruritus (General disorders) | 0 (0) | 1 (1)
Catheter Site Rash (General disorders) | 1 (1) | 1 (1)
Catheter Site Related Reaction (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 7 (7)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Feeling Jittery (General disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 9 (9) | 3 (3)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 13 (13) | 10 (10)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Implant Site Infection (Infections and infestations) | 1 (1) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion Site Vesicles (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 2 (2) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Medical Device Complication (General disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscloskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (10) | 7 (7)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 15 (15) | 10 (10)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal Failure Acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Tropinin Increased (Investigations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vulvovaginal Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The EPITOME-1 study is an open label study without a primary endpoint. The sample size was determined based on feasibility and not a power calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No